CLINICAL TRIAL: NCT02084537
Title: Minimally Invasive Surgery vs. Endoscopy Randomized (MISER) Trial for Necrotizing Pancreatitis
Acronym: MISER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 577235
Record Dates: First submitted 2014-03-10; First posted 2014-03-12 (Estimated); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Necrosis of Pancreas; Infected Pancreatic Necrosis
Keywords: symptomatic; infected; necrotic collection
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endoscopic treatment (Active Comparator): Treated by single or multiple transmural cystogastrostomy tracts, 15mm balloon dilation, two 7 French (Fr) double pigtail plastic stents or lumen-apposing metal stents and nasocystic drainage catheter, with or without endoscopic necrosectomy as needed.
  Interventions: Procedure: Endoscopic treatment
- Minimally invasive surgical necrosectomy (Active Comparator): Video-assisted retroperitoneal debridement (VARD) or laparoscopic approach. This includes laparoscopic cystogastrostomy with internal debridement.
  Interventions: Procedure: Minimally invasive surgical necrosectomy

INTERVENTIONS:
Procedure: Endoscopic treatment — Treated by single or multiple transmural cystogastrostomy tracts, 15mm balloon dilation, two 7fr double pigtail plastic stents or lumen-apposing metal stents and nasocystic drainage catheter, with or without endoscopic necrosectomy as needed.
  Other Names: Endoscopic cystogastrostomy; Endoscopic cystoduodenostomy; Endoscopic necrosectomy
  Arms: Endoscopic treatment
Procedure: Minimally invasive surgical necrosectomy — Video-assisted retroperitoneal debridement (VARD) or laparoscopic cystogastrostomy with internal debridement.
  Other Names: Video-assisted retroperitoneal debridement (VARD); Laparoscopic cystogastrostomy with internal debridement
  Arms: Minimally invasive surgical necrosectomy

SUMMARY:
Prospective, randomized controlled trial comparing Endoscopic Ultrasound (EUS) Guided cystogastrostomy or cystoduodenostomy and endoscopic necrosectomy to minimally invasive surgical necrosectomy, in patients with necrotizing pancreatitis.

DETAILED DESCRIPTION:
Patients will be randomly allocated to either treatment arm in a 1:1 ratio. Following intervention, patients will be assessed at regular intervals until study completion at 6 months post-discharge. Primary outcome is a composite of major complications and/or mortality, measured to 6 months post-discharge.

ELIGIBILITY:
Inclusion Criteria:

* Necrotic collection

  * Infected (suspected and confirmed): clinical signs of infection (septic, positive cultures, febrile), systemic inflammatory response syndrome, gas within the collection on imaging (not iatrogenic), or positive culture of collection contents
* Necrotic collection is within 15mm of the lumen of the gastrointestinal tract.
* 18 years and older
* Informed consent obtained from the patient or their medical representative.
* Medically fit for general anesthetic
* Collection amenable to either endoscopic or minimally invasive surgical necrosectomy and drainage.

Exclusion Criteria:

* <18 years old
* Unable to obtain informed consent from the patient or their medical representative.
* Medically unfit for general anesthesia
* Pregnant
* Necrotic collection not accessible by either or both techniques
* The collection is >15mm from the lumen of the gastrointestinal tract.
* Irreversible coagulopathy: International Normalized Ratio (INR) >1.5
* Irreversible thrombocytopenia: platelet count <50 x10^9/L
* Dual antiplatelet therapy or therapeutic anticoagulation that cannot be withheld for the procedure
* Surgical or endoscopic necrosectomy or pseudocyst drainage has been performed within the preceding 12 months
* Necrotic collection secondary to trauma or other surgical event that requires additional interventions such as management of liver lacerations or vascular injury.
* Pre-existing percutaneous drain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2014-04; Primary Completion 2017-12-31 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Major complications | 6 months post discharge
  Composite of major complications and/or mortality (all cause and disease specific), measured to 6 months post discharge

CONTACTS AND LOCATIONS:
Overall Officials: Shyam S Varadarajulu, MD, Principal Investigator — AdventHealth
Locations (1):
- Florida Hospital Center for Interventional Endoscopy, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bang JY, Arnoletti JP, Holt BA, Sutton B, Hasan MK, Navaneethan U, Feranec N, Wilcox CM, Tharian B, Hawes RH, Varadarajulu S. An Endoscopic Transluminal Approach, Compared With Minimally Invasive Surgery, Reduces Complications and Costs for Patients With Necrotizing Pancreatitis. Gastroenterology. 2019 Mar;156(4):1027-1040.e3. doi: 10.1053/j.gastro.2018.11.031. Epub 2018 Nov 16. PMID 30452918